CLINICAL TRIAL: NCT02180867
Title: Pazopanib Neoadjuvant Trial in Non-Rhabdomyosarcoma Soft Tissue Sarcomas (PAZNTIS): A Phase II/III Randomized Trial of Preoperative Chemoradiation or Preoperative Radiation Plus or Minus Pazopanib (NSC# 737754)
Brief Title: Radiation Therapy With or Without Combination Chemotherapy or Pazopanib Before Surgery in Treating Patients With Newly Diagnosed Non-rhabdomyosarcoma Soft Tissue Sarcomas That Can Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01340; NCI-2014-01340 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ARST1321; s14-02023; ARST1321 (Other: Children's Oncology Group); ARST1321 (Other: CTEP); U10CA098543 (NIH); U10CA180830 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Alveolar Soft Part Sarcoma; Angiomatoid Fibrous Histiocytoma; Atypical Fibroxanthoma; Clear Cell Sarcoma of Soft Tissue; Epithelioid Malignant Peripheral Nerve Sheath Tumor; Epithelioid Sarcoma; Extraskeletal Myxoid Chondrosarcoma; Extraskeletal Osteosarcoma; Fibrohistiocytic Neoplasm; Fibrosarcoma; Inflammatory Myofibroblastic Tumor; Intimal Sarcoma; Leiomyosarcoma; Liposarcoma; Liver Embryonal Sarcoma; Low Grade Fibromyxoid Sarcoma; Low Grade Myofibroblastic Sarcoma; Malignant Peripheral Nerve Sheath Tumor; Malignant Skin Granular Cell Tumor; Malignant Triton Tumor; Mesenchymal Chondrosarcoma; Myxofibrosarcoma; Myxoid Chondrosarcoma; Myxoinflammatory Fibroblastic Sarcoma; Nerve Sheath Neoplasm; PEComa; Pericytic Neoplasm; Plexiform Fibrohistiocytic Tumor; Sclerosing Epithelioid Fibrosarcoma; Skin Glomus Tumor; Stage IB Soft Tissue Sarcoma AJCC v7; Stage IIB Soft Tissue Sarcoma AJCC v7; Stage III Soft Tissue Sarcoma AJCC v7; Stage IV Soft Tissue Sarcoma AJCC v7; Synovial Sarcoma; Undifferentiated High Grade Pleomorphic Sarcoma of Bone
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Histiocytoma, Angiomatoid Fibrous; Sarcoma, Clear Cell; Sarcoma; Chondrosarcoma, Extraskeletal Myxoid; Fibrosarcoma; Granuloma, Plasma Cell; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Chondrosarcoma, Mesenchymal; Dermatofibrosarcoma; Nerve Sheath Neoplasms; Perivascular Epithelioid Cell Neoplasms; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous | interventions — Doxorubicin; Ifosfamide; pazopanib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regimen A (pazopanib, chemoradiation) (Experimental): See Regimen A Detailed Description.
  Interventions: Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Ifosfamide; Drug: Pazopanib; Drug: Pazopanib Hydrochloride; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery
- Regimen B (chemoradiation) (Experimental): See Regimen B Detailed Description.
  Interventions: Drug: Doxorubicin; Drug: Doxorubicin Hydrochloride; Drug: Ifosfamide; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery
- Regimen C (pazopanib, radiation therapy) (Experimental): INDUCTION PHASE: Patients receive pazopanib PO QD on weeks 1-9. Patients undergo radiation therapy on weeks 1-7.
  SURGERY: Patients undergo surgery on week 10.
  CONTINUATION PHASE: Patients receive pazopanib PO QD on weeks 13-25. If applicable, patients undergo additional radiation therapy at week 13.
  Interventions: Drug: Pazopanib; Drug: Pazopanib Hydrochloride; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery
- Regimen D (radiation therapy) (Experimental): INDUCTION PHASE: Patients undergo radiation therapy on weeks 1-7.
  SURGERY: Patients undergo surgery on week 10.
  CONTINUATION PHASE: If applicable, patients undergo additional radiation therapy at week 13.
  Interventions: Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Regimen A (pazopanib, chemoradiation); Regimen B (chemoradiation)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
  Arms: Regimen A (pazopanib, chemoradiation); Regimen B (chemoradiation)
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
  Arms: Regimen A (pazopanib, chemoradiation); Regimen B (chemoradiation)
Drug: Pazopanib — Given PO
  Other Names: GW786034
  Arms: Regimen A (pazopanib, chemoradiation); Regimen C (pazopanib, radiation therapy)
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW 786034B; GW-786034B; GW786034B; Pazopater; Votrient
  Arms: Regimen A (pazopanib, chemoradiation); Regimen C (pazopanib, radiation therapy)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This randomized phase II/III trial studies how well pazopanib, when combined with chemotherapy and radiation therapy or radiation therapy alone, work in the treatment of patients with newly diagnosed non-rhabdomyosarcoma soft tissue sarcomas that can eventually be removed by surgery. Radiation therapy uses high energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as ifosfamide and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Pazopanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether these therapies can be safely combined and if they work better when given together in treating patients with non-rhabdomyosarcoma soft tissue sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the dose of pazopanib that is feasible when given in combination with radiation or chemoradiation in pediatric and adult patients newly diagnosed with unresected intermediate- and high-risk non rhabdomyosarcoma soft tissue sarcomas (NRSTS).

II. To compare the rates of near complete pathologic response (> 90% necrosis) with the addition of pazopanib to preoperative chemoradiation versus preoperative chemoradiation alone for potentially resectable > 5 cm, grade 2 or 3 intermediate to high risk chemotherapy-sensitive NRSTS in the phase II portion of the study for this cohort.

III. To compare the rates of near complete pathologic response (> 90% necrosis) with the addition of pazopanib to preoperative radiotherapy versus preoperative radiotherapy alone for potentially resectable intermediate to high risk adult and pediatric NRSTS in the phase II portion of the study for this cohort (using a phase II decision rule to go onto the phase III portion of the study).

IV. To compare the rates of event-free survival (EFS) with the addition of pazopanib to preoperative radiotherapy versus preoperative radiotherapy alone for localized intermediate to high risk adult and pediatric NRSTS in the phase III portion of the study for this cohort if the phase II decision rule is passed.

SECONDARY OBJECTIVES:

I. To estimate the rates of local failure, regional failure, distant metastasis free survival, disease-free survival, and overall survival with the addition of pazopanib to preoperative chemoradiation or preoperative radiation in intermediate to high risk adult and pediatric NRSTS.

II. To compare the pattern of recurrence (local, regional and distant) between preoperative chemoradiation or radiation with the addition of pazopanib for adult and pediatric NRSTS.

III. To define the toxicities of ifosfamide and doxorubicin chemotherapy and radiation when used in combination with pazopanib in intermediate to high risk adult and pediatric NRSTS.

IV. To define the toxicities of preoperative radiotherapy when used in combination with pazopanib in intermediate to high risk adult and pediatric NRSTS.

EXPLORATORY OBJECTIVES:

I. To gain insight into the disease biology of childhood and adult NRSTS through analysis of actionable mutations and whole genome sequencing.

II. To determine if microvessel density and circulating tumor deoxyribonucleic acid (DNA) predict response to pazopanib and outcome.

III. To determine the effect of pazopanib on doxorubicin exposure in children and adults with NRSTS.

IV. To evaluate change in fludeoxyglucose F 18 (FDG) positron emission tomography (PET) maximum standard uptake value (SUVmax) from baseline to week 10 or 13 in patients with unresected tumors and to correlate this change with pathologic response and EFS.

V. To compare the rate of response by standard imaging and pathologic assessment to determine which correlates better with local tumor control, distant tumor control, EFS, and overall survival.

OUTLINE: This study starts as a dose-escalation study of pazopanib.

CHEMOTHERAPY COHORT: Patients eligible for chemotherapy cohort are randomized to 1 of 2 treatment regimens.

REGIMEN A:

INDUCTION PHASE: Patients receive pazopanib orally (PO) once daily (QD) on weeks 1-12, ifosfamide intravenously (IV) over 2-4 hours on days 1-3 on weeks 1, 4, 7, 10, and doxorubicin IV over 1-15 minutes on days 1-2 on weeks 1 and 4. At least 24 hours after the completion of week 4 doxorubicin, patients undergo radiation therapy on weeks 4-10.

SURGERY: Patients undergo surgery on week 13.

CONTINUATION PHASE: Patients receive pazopanib PO QD on weeks 16-25, ifosfamide IV over 2-4 hours on days 1-3 on weeks 16 and 19, and doxorubicin IV over 1-15 minutes on days 1-2 on weeks 16, 19, and 22. If applicable, patients undergo additional radiation therapy at week 16

REGIMEN B:

INDUCTION PHASE: Patients receive ifosfamide IV over 2-4 hours on days 1-3 on weeks 1, 4, 7, 10 and doxorubicin hydrochloride IV over 1-15 minutes on days 1-2 on weeks 1 and 4. At least 24 hours after the completion of week 4 doxorubicin, patients undergo radiation therapy on weeks 4-10.

SURGERY: Patients undergo surgery on week 13.

CONTINUATION PHASE: Patients receive ifosfamide IV over 2-4 hours on days 1-3 on weeks 16 and 19 and doxorubicin IV over 1-15 minutes on days 1-2 on weeks 16, 19, and 22. If applicable, patients undergo additional radiation therapy at week 16.

NON-CHEMOTHERAPY COHORT: Patients eligible for non-chemotherapy cohort are randomized to 1 of 2 treatment regimens.

REGIMEN C:

INDUCTION PHASE: Patients receive pazopanib PO QD on weeks 1-9. Patients undergo radiation therapy on weeks 1-7.

SURGERY: Patients undergo surgery on week 10.

CONTINUATION PHASE: Patients receive pazopanib PO QD on weeks 13-25. If applicable, patients undergo additional radiation therapy at week 13.

REGIMEN D:

INDUCTION PHASE: Patients undergo radiation therapy on weeks 1-7.

SURGERY: Patients undergo surgery on week 10.

CONTINUATION PHASE: If applicable, patients undergo additional radiation therapy at week 13.

After completion of study treatment, patients are followed up at 6, 12, 18, 24, 30, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Note: eligible patients must have a body surface area >= 0.5 m^2 AND be able to swallow whole tablets
* Newly diagnosed and histopathologically confirmed, potentially resectable NRSTS of the extremity and trunk will be eligible for the chemotherapy or non-chemotherapy cohort based on:

  * Evidence of chemotherapy sensitivity of the histologic sarcoma subtype based on existing evidence from prior clinical trials
  * Sufficient risk of metastatic disease to warrant chemotherapy based on size and grade and
  * Medically deemed able or unable to undergo chemotherapy
  * Notes: an incisional biopsy or core biopsy is preferred; fine needle aspiration biopsy is not acceptable to establish the diagnosis
* ELIGIBLE SITES:

  * Extremities: upper (including shoulder) and lower (including hip)
  * Trunk: body wall
* INELIGIBLE SITES: Head and neck, visceral organs (with the exception of embryonal sarcoma of the liver), retroperitoneum, peritoneum, pelvis within the confines of the bony pelvis
* ELIGIBILITY FOR CHEMOTHERAPY COHORT:
* Stage T2a/b (> 5 cm) and grade 2 or 3 AND
* One of the following chemosensitive histologies as defined in the World Health Organization (WHO) classification of soft tissue tumors (with some evidence of good response to chemoradiation and of sufficient high risk of metastases, or clear evidence of metastases):

  * Unclassified soft tissue sarcomas that are too undifferentiated to be placed in a specific pathologic category in the WHO classification (often called "undifferentiated soft tissue sarcoma" or "soft tissue sarcoma not otherwise specified [NOS]")
  * Synovial sarcoma
  * Angiosarcoma of soft tissue
  * Adult fibrosarcoma
  * Mesenchymal (extraskeletal) chondrosarcoma
  * Leiomyosarcoma
  * Liposarcoma (excluding myxoid liposarcoma)
  * Undifferentiated pleomorphic sarcoma
  * Embryonal sarcoma of the liver
* Patients meeting the above criteria (histology, size, and grade) with the EXCEPTION of histologies noted above may enroll on the chemotherapy cohort or the non-chemotherapy cohort at the discretion of the enrolling investigator; patients meeting these criteria with the EXCEPTION of histologies noted above but medically deemed unable to receive chemotherapy or who elect not to receive chemotherapy are eligible for the non-chemotherapy cohort
* Patients with the following histologies are only eligible for the chemotherapy cohort and cannot enroll on the non-chemotherapy cohort:

  * Unclassified soft tissue sarcomas that are too undifferentiated to be placed in a specific pathologic category in the WHO classification (often called "undifferentiated soft tissue sarcoma" or "soft tissue sarcoma NOS") in patients < 30 years of age
  * Synovial sarcoma
  * Embryonal sarcoma of the liver
* ELIGIBILITY FOR NON-CHEMOTHERAPY COHORT:
* Patients with any size of grade 2 or 3 of the following "intermediate (rarely metastasizing)" or "malignant" tumors, as defined in the WHO classification of soft tissue tumors for which we have consensus data of chemotherapy-resistance are eligible only for the non-chemotherapy cohort:

  * So-called fibrohistiocytic tumors - plexiform fibrohistiocytic tumor, giant cell tumor of soft tissues
  * Fibroblastic/myofibroblastic tumors - solitary fibrous tumor, malignant solitary fibrous tumor, inflammatory myofibroblastic tumor, low grade myofibroblastic sarcoma, myxoinflammatory fibroblastic sarcoma, atypical myxoinflammatory fibroblastic tumor, myxofibrosarcoma, low grade fibromyxoid sarcoma, sclerosing epithelioid fibrosarcoma
  * Tumors of uncertain differentiation - epithelioid sarcoma, alveolar soft part sarcoma, clear cell sarcoma of soft tissue, angiomatoid fibrous histiocytoma, ossifying fibromyxoid tumor, myoepithelioma, myoepithelial carcinoma, extraskeletal myxoid chondrosarcoma, neoplasms with perivascular epithelioid cell differentiation (PEComa), intimal sarcoma, atypical fibroxanthoma, mixed tumor NOS, phosphaturic mesenchymal tumor, malignant ossifying fibromyxoid tumor, malignant mixed tumor, malignant phosphaturic mesenchymal tumor
  * Chondro-osseous tumors - extraskeletal osteosarcoma
  * Pericytic (perivascular) tumors - malignant glomus tumor
  * Nerve sheath tumors - malignant peripheral nerve sheath tumor, malignant granular cell tumor, epithelioid malignant peripheral nerve sheath tumor, malignant Triton tumor
  * Undifferentiated sarcomas (with a specific pathologic category in the WHO classification) - undifferentiated round cell sarcoma, undifferentiated epithelioid sarcoma, undifferentiated spindle cell sarcoma
* Patients meeting the criteria (histology, size, and grade) with the EXCEPTION of histologies noted above may enroll on the non-chemotherapy cohort at the discretion of the enrolling investigator; patients meeting these criteria with the EXCEPTION of histologies noted above but medically deemed unable to receive chemotherapy or who elect not to receive chemotherapy are eligible for the non-chemotherapy cohort; note that tumors arising in bone are NOT eligible for this study
* Extent of disease:

  * Patients with non-metastatic and metastatic disease are eligible
  * Initially unresectable patients, with or without metastatic disease, are eligible as long as there is a commitment at enrollment to resect the primary tumor
* Sufficient tissue and blood must be available to submit for required biology studies
* Lansky performance status score >= 70 for patients =< 16 years of age
* Karnofsky performance status score >= 70 for patients > 16 years of age
* Absolute neutrophil count >= 1500/uL; Note: no transfusions are permitted 7 days prior to laboratory studies to determine eligibility
* Platelet count >= 100,000/uL; Note: no transfusions are permitted 7 days prior to laboratory studies to determine eligibility
* Hemoglobin >= 8 g/dL for patients =< 16 years of age; >= 9 g/dL for patients > 16 years of age; Note: no transfusions are permitted 7 days prior to laboratory studies to determine eligibility
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or normal serum creatinine based on age/gender as follows:

  * 2 to < 6 years; 0.8 mg/dL male; 0.8 mg/dL female
  * 6 to < 10 years; 1 mg/dL male; 1 mg/dL female
  * 10 to < 13 years; 1.2 mg/dL male; 1.2 mg/dL female
  * 13 to < 16 years; 1.5 mg/dL male; 1.4 mg/dL female
  * >= 16 years; 1.5 mg/dL male; 1.4 mg/dL female
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 2.5 x upper limit of normal (ULN) for age
* Shortening fraction of >= 27% by echocardiogram OR ejection fraction of >= 50% by radionuclide angiogram
* Corrected QT interval (QTc) < 480 msec
* No evidence of dyspnea at rest, no exercise intolerance, and a resting pulse oximetry reading > 94% on room air if there is clinical indication for determination
* Patients on low molecular weight heparin or Coumadin (with a stable international normalized ratio [INR]) are eligible
* Patient must have a life expectancy of at least 3 months with appropriate therapy
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients with grade 1 NRSTS tumors of any size are not eligible
* Patients with known central nervous system (CNS) metastases are not eligible; Note: brain imaging is not an eligibility requirement
* Patients with evidence of active bleeding or bleeding diathesis will be excluded (Note: patients aged > 17 years with excess of 2.5 mL of hemoptysis are not eligible)
* Patients with gross total resection of the primary tumor prior to enrollment on ARST1321 are NOT eligible; patients who have experienced tumor recurrence after a gross total tumor resection are NOT eligible
* Patients with uncontrolled hypertension are ineligible; uncontrolled hypertension is defined as follows:

  * Patients aged =< 17 years: greater than 95th percentile systolic and diastolic blood pressure based on age and height which is not controlled by one anti-hypertensive medication
  * Patients aged > 17 years: systolic blood pressure >= 140 mmHg and/or diastolic blood pressure >= 90 mmHg that is not controlled by one anti-hypertensive medication
* Prior Therapy:

  * Patients must have had no prior anthracycline (e.g., doxorubicin, daunorubicin) or ifosfamide chemotherapy
  * Patients must have had no prior use of pazopanib or similar multi-targeted tyrosine kinase inhibitors (TKI)
  * Patients must have had no prior radiotherapy to tumor-involved sites
  * Note: patients previously treated for a non-NRSTS cancer are eligible provided they meet the prior therapy requirements; patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are excluded
* Other types of invasive malignancy that are not disease free within 3 years except for non-melanoma skin cancer, lentigo maligna, any carcinoma-in-situ or prostate cancer with low risk factors
* CYTOCHROME P450 3A4 (CYP3A4) substrates WITH narrow therapeutic indices: patients chronically receiving medications known to be metabolized by CYP3A4 and with narrow therapeutic indices within 7 days prior to study enrollment, including but not limited to pimozide, aripiprazole, triazolam, ergotamine and halofantrine are not eligible; Note: the use of fentanyl is permitted
* CYP3A4 Inhibitors: patients chronically receiving drugs that are known potent CYP3A4 inhibitors within 7 days prior to study enrollment, including but not limited to itraconazole, clarithromycin, erythromycin many non-nucleoside reverse-transcriptase inhibitors (NNRTIs), diltiazem, verapamil, and grapefruit juice are not eligible
* CYP3A4 Inducers: patients chronically receiving drugs that are known potent CYP3A4 inducers within 14 days prior to study enrollment, including but not limited to carbamazepine, phenobarbital, phenytoin, rifampin, and St. John's wort are not eligible (with the exception of glucocorticoids)
* Certain medications that are associated with a risk for QTc prolongation and/or Torsades de Pointes, although not prohibited, should be avoided or replaced with medications that do not carry these risks, if possible
* Subjects with any condition that may impair the ability to swallow or absorb oral medications/investigational product including:

  * Any lesion, whether induced by tumor, radiation or other conditions, which makes it difficult to swallow capsules or pills
  * Prior surgical procedures affecting absorption including, but not limited to major resection of stomach or small bowel
  * Active peptic ulcer disease
  * Malabsorption syndrome
* Subjects with any condition that may increase the risk of gastrointestinal bleeding or gastrointestinal perforation, including:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesions
  * Inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease) or other gastrointestinal conditions which increase the risk of perforation
  * History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 28 days prior to beginning study treatment
* Subjects with any of the following cardiovascular conditions within the past 6 months

  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Cardiac arrhythmia
  * Admission for unstable angina
  * Cardiac angioplasty or stenting
  * Coronary artery bypass graft surgery
  * Pulmonary embolism, untreated deep venous thrombosis (DVT) or DVT which has been treated with therapeutic anticoagulation for less than 6 weeks
  * Arterial thrombosis
  * Symptomatic peripheral vascular disease
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; a subject who has a history of class II heart failure and is asymptomatic on treatment may be considered eligible
* History of serious or non-healing wound, ulcer, or bone fracture
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are unable to swallow whole tablets are not eligible
* Patients with a body surface area < 0.5 m^2 are not eligible
* Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with pazopanib; in addition, these subjects are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Patients who are receiving any other investigational agent(s)
* Pregnancy and breast feeding:

  * Female patients who are pregnant are ineligible due to risks of fetal and teratogenic adverse events as seen in animal/human studies
  * Lactating females are not eligible unless they have agreed not to breastfeed their infants during treatment and for a period of 1 month following completion of treatment
  * Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Unwillingness to use an effective contraceptive method for the duration of their study participation and for at least 1 month after treatment is completed if sexually active with reproductive potential

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-07-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2025-12-23 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron R Weiss, Principal Investigator — Children's Oncology Group
Locations (381):
- United States (365):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Children's Hospital Colorado, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Saint John's Hospital, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Newman Regional Health, Emporia, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Drexel University School of Medicine, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Canada (14):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Puerto Rico (2):
  - San Jorge Children's Hospital, San Juan
  - University Pediatric Hospital, San Juan

REFERENCES:
- [Derived] Weiss AR, Chen YL, Scharschmidt TJ, Xue W, Gao Z, Black JO, Choy E, Davis JL, Fanburg-Smith JC, Kao SC, Kayton ML, Kessel S, Lim R, Million L, Okuno SH, Ostrenga A, Parisi MT, Pryma DA, Randall RL, Rosen MA, Shulkin BL, Terezakis S, Venkatramani R, Zambrano E, Wang D, Hawkins DS, Spunt SL. Outcomes After Preoperative Chemoradiation With or Without Pazopanib in Non-Rhabdomyosarcoma Soft Tissue Sarcoma: A Report From Children's Oncology Group and NRG Oncology. J Clin Oncol. 2023 Nov 1;41(31):4842-4848. doi: 10.1200/JCO.23.00045. Epub 2023 Jul 31. PMID 37523624
- [Derived] Avutu V, Weiss AR, Reed DR, Ahmed SK, Allen-Rhoades WA, Chen YE, Davis LE, Eaton BR, Hawkins DS, Indelicato DJ, Patel SR, Randall RL, Reinke DK, Riedel RF, Scharschmidt TJ, Thornton KA, Wang D, Janeway KA, Kopp LM. Identified Enrollment Challenges of Adolescent and Young Adult Patients on the Nonchemotherapy Arm of Children's Oncology Group Study ARST1321. J Adolesc Young Adult Oncol. 2022 Jun;11(3):328-332. doi: 10.1089/jayao.2021.0103. Epub 2021 Sep 9. PMID 34515544
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353
- [Derived] Weiss AR, Chen YL, Scharschmidt TJ, Chi YY, Tian J, Black JO, Davis JL, Fanburg-Smith JC, Zambrano E, Anderson J, Arens R, Binitie O, Choy E, Davis JW, Hayes-Jordan A, Kao SC, Kayton ML, Kessel S, Lim R, Meyer WH, Million L, Okuno SH, Ostrenga A, Parisi MT, Pryma DA, Randall RL, Rosen MA, Schlapkohl M, Shulkin BL, Smith EA, Sorger JI, Terezakis S, Hawkins DS, Spunt SL, Wang D. Pathological response in children and adults with large unresected intermediate-grade or high-grade soft tissue sarcoma receiving preoperative chemoradiotherapy with or without pazopanib (ARST1321): a multicentre, randomised, open-label, phase 2 trial. Lancet Oncol. 2020 Aug;21(8):1110-1122. doi: 10.1016/S1470-2045(20)30325-9. Epub 2020 Jul 20. PMID 32702309

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients began at Dose-Finding Level 1. Dose-Finding Level 0 CR, Dose-Finding Level 2 CR, and Dose-Finding Level 0 RT never enrolled because protocol-defined dose de-escalation and escalation parameters were not met. Cohorts C and D were closed to further patient accrual on October 12, 2017 due to slower than anticipated enrollment.
Groups:
- Dose-Finding Level 1 CR: Dose-Finding Level 1 CR:
  Adult: Pazopanib 600 mg; Pediatric: Pazopanib 350 mg/m2
- Dose-Finding Level 1 RT: Dose-Finding Level 1 RT:
  Adult: Pazopanib 600 mg; Pediatric: Pazopanib 350 mg/m2
- Dose-Finding Level 2 RT: Dose-Finding Level 2 RT:
  Adult: Pazopanib 800 mg; Pediatric: Pazopanib 450 mg/m2
- Regimen A: Regimen A: Chemoradiation plus pazopanib
- Regimen B: Regimen B: Chemoradiation alone
- Regimen C: Regimen C: Radiation therapy plus pazopanib
- Regimen D: Regimen D: Radiation therapy alone
Period: Overall Study
Arm/Group | Dose-Finding Level 1 CR | Dose-Finding Level 1 RT | Dose-Finding Level 2 RT | Regimen A | Regimen B | Regimen C | Regimen D
Started | 10 | 11 | 10 | 49 | 48 | 6 | 6
Pediatric Patients | 6 | 4 | 3 | 18 | 19 | 1 | 0
Adult Patients | 4 | 7 | 7 | 31 | 29 | 5 | 6
Completed | 4 | 0 | 6 | 23 | 21 | 3 | 1
Not Completed | 6 | 11 | 4 | 26 | 27 | 3 | 5
Not completed — Adverse Event | 3 | 4 | 1 | 5 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 1 | 6 | 0 | 1
Not completed — Physician Decision | 1 | 3 | 1 | 10 | 9 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Ineligible | 1 | 2 | 0 | 3 | 5 | 0 | 0
Not completed — Repeat Eligibility Studies | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Refusal of further protocol therapy | 1 | 0 | 2 | 6 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: It was pre-specified to combine adult and pediatric participants for analysis as they received an equivalent dose of Pazopanib. There were no patients enrolled onto Dose-Finding Level 0 CR and Dose-Finding Level 2 CR or Dose-Finding Level 0 RT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-Finding Level 1 CR | Dose-Finding Level 1 RT | Dose-Finding Level 2 RT | Regimen A | Regimen B | Regimen C | Regimen D | Total
Number analyzed (Participants) | 10 | 11 | 10 | 49 | 48 | 6 | 6 | 140
Age, Continuous [Mean (Standard Deviation); unit: Months] | 225.1 (57.8) | 524.3 (270.3) | 407.3 (224.7) | 376.3 (243.4) | 356.2 (221.8) | 547.2 (260.6) | 722.8 (141.9) | 394.6 (242.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 30 | 18 | 2 | 3 | 63
  Male | 6 | 8 | 7 | 19 | 30 | 4 | 3 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 13 | 9 | 0 | 0 | 26
  Not Hispanic or Latino | 6 | 9 | 9 | 34 | 38 | 6 | 6 | 108
  Unknown or Not Reported | 2 | 1 | 0 | 2 | 1 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 3 | 6 | 1 | 0 | 15
  White | 7 | 8 | 8 | 39 | 38 | 5 | 5 | 110
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 7 | 3 | 0 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Feasible Dose: Pediatric
Description: The dose of pazopanib that is feasible when given in combination with radiation or chemoradiation in pediatric unresected intermediate- and high-risk NRSTS patients. Initially, up to 10 patients (minimum of 3 patients ≥ 2 and < 18 years of age and 3 patients ≥ 18 years of age) eligible for each of the two study cohorts were non-randomly assigned (to generate 8 patients evaluable for toxicity) to receive treatment with pazopanib at dose level 1. A protocol-defined list of pazopanib-associated adverse events were defined as dose-limiting toxicities. The pazopanib dose determined to be feasible was based on the number of patient-reported dose-limiting toxicities encountered.
Time Frame: After the first 6 weeks of Induction
Population: Pediatric patients, excluding 1 ineligible patient in Dose-Finding CR group and 1 ineligible patient in Dose-Finding RT group
Measure: Number; unit: milligram per square meter
Groups:
- All Pediatric Dose Finding CR Cohorts: Dose-Finding CR: Chemoradiation plus pazopanib
- All Pediatric Dose Finding RT Cohorts: Dose-Finding RT: Radiation therapy plus pazopanib
Arm/Group | All Pediatric Dose Finding CR Cohorts | All Pediatric Dose Finding RT Cohorts
Number analyzed (Participants) | 5 | 6
milligram per square meter | 350 | 450

2. Primary Outcome: Feasible Dose: Adult
Description: The dose of pazopanib that is feasible when given in combination with radiation or chemoradiation in adult unresected intermediate- and high-risk NRSTS patients. Initially, up to 10 patients (minimum of 3 patients ≥ 2 and < 18 years of age and 3 patients ≥ 18 years of age) eligible for each of the two study cohorts were non-randomly assigned (to generate 8 patients evaluable for toxicity) to receive treatment with pazopanib at dose level 1. A protocol-defined list of pazopanib-associated adverse events were defined as dose-limiting toxicities. The pazopanib dose determined to be feasible was based on the number of patient-reported dose-limiting toxicities encountered.
Time Frame: After the first 6 weeks of Induction
Population: Adult patients, excluding 1 ineligible patient in Dose-Finding RT group
Measure: Number; unit: milligram
Groups:
- All Adult Dose Finding CR Cohorts: Dose-Finding CR: Chemoradiation plus pazopanib
- All Adult Dose Finding RT Cohorts: Dose-Finding RT: Radiation therapy plus pazopanib
Arm/Group | All Adult Dose Finding CR Cohorts | All Adult Dose Finding RT Cohorts
Number analyzed (Participants) | 4 | 13
milligram | 600 | 800

3. Primary Outcome: Percentage of Chemoradiotherapy Patients With Positive Pathologic Response at Week 13
Description: A responder is defined by more than (90% tumor necrosis at week 13). A non-responder has less than 90% necrosis or progressive disease before week 13.
Time Frame: Week 13 after induction
Population: It was pre-specified to combine adult and pediatric participants for analysis as they received an equivalent dose of Pazopanib. There were no patients enrolled onto Dose-Finding Level 0 CR or Dose-Finding Level 2 CR. 19 Regimen A patients and 23 Regimen B patients were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Dose-Finding Level 1 CR | Regimen A | Regimen B
Number analyzed (Participants) | 6 | 30 | 25
Percentage of patients | 66.67 [28.95 to 100] | 46.67 [28.81 to 64.52] | 24 [7.26 to 40.74]

4. Primary Outcome: Percentage of Radiotherapy Patients With Positive Pathologic Response at Week 10
Description: A responder is defined by more than 90% tumor necrosis at week 10. A non-responder has less than 90% necrosis or progressive disease before week 10.
Time Frame: Week 10 after induction
Population: It was pre-specified to combine adult and pediatric participants for analysis as they received an equivalent dose of Pazopanib. There were no patients enrolled onto Dose Level 0 RT. 3 Regimen C patients excluded: 1 patient did not receive treatment and 2 missing review; 4 Regimen D patients excluded due to missing review.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Dose-Finding Level 1 RT | Dose-Finding Level 2 RT | Regimen C | Regimen D
Number analyzed (Participants) | 3 | 5 | 3 | 2
Percentage of patients | 0 [0 to 0] | 40 [0 to 82.94] | 0 [0 to 0] | 0 [0 to 0]

5. Primary Outcome: Percentage of Radiotherapy Patients Failure Free at 5 Years Following Study Entry
Description: Time to the first occurrence of relapse, progression, secondary cancer or death from any cause.
Time Frame: From enrollment to up to 60 months
Population: Data for the phase III portion of the study were never collected because the RT arm was closed earlier due to slow accrual.
Arm/Group | Regimen C | Regimen D
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Patients Local Failure Free at 5 Years Following Study Entry
Description: Defined as disease recurrence only at the primary site of disease at diagnosis. The relative risk of specific failure types will be estimated and compared descriptively using the Cox proportional hazard model. Data were obtained from institutional reported data.
Time Frame: From enrollment to up to 60 months
Population: Patients deemed ineligible in the original cohort are excluded. An additional five (5) patients are excluded in this 5-year analysis as they were deemed ineligible post the initial submission and publication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Finding Level 1 CR | Dose-Finding Level 1 RT | Dose-Finding Level 2 RT | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 9 | 9 | 10 | 44 | 41 | 5 | 6
percentage of participants | 100.00 [100.00 to 100.00] | 80.00 [30.42 to 100.00] | 100.00 [100.00 to 100.00] | 91.09 [77.33 to 100.00] | 87.32 [68.05 to 100.00] | 100.00 [100.00 to 100.00] | 83.33 [16.65 to 100.00]

7. Secondary Outcome: Percentage of Patients Regional Failure Free at 5 Years Following Study Entry
Description: Defined as disease recurrence at lymph nodes regional to the primary disease site, with or without local failure but without distant failure. The relative risk of specific failure types will be estimated and compared descriptively using the Cox proportional hazard model. Data were obtained from institutional reported data.
Time Frame: From enrollment to up to 60 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Finding Level 1 CR | Dose-Finding Level 1 RT | Dose-Finding Level 2 RT | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 9 | 9 | 10 | 44 | 41 | 5 | 6
percentage of participants | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00] | 100.00 [100.00 to 100.00]

8. Secondary Outcome: Percentage of Patients Distant Failure Free at 5 Years Following Study Entry
Description: Defined as disease recurrence at sites other than the primary site and diagnosis and nodes regional to that site (metastatic disease, whether or not present at diagnosis), with or without loco-regional failure. The relative risk of specific failure types will be estimated and compared descriptively using the Cox proportional hazard model. Data were obtained from institutional reported data.
Time Frame: From enrollment to up to 60 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-Finding Level 1 CR | Dose-Finding Level 1 RT | Dose-Finding Level 2 RT | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 9 | 9 | 10 | 44 | 41 | 5 | 6
percentage of participants | 77.78 [48.44 to 100.00] | 33.33 [0.00 to 71.05] | 70.00 [32.43 to 100.00] | 59.89 [39.11 to 78.67] | 62.62 [39.99 to 85.24] | 80.00 [39.52 to 100.00] | 66.67 [0.00 to 100.00]

9. Secondary Outcome: Percentage of Patients Who Experienced Grade 3 or Higher Toxicity Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Description: Participants who experienced Grade 3 or higher toxicity was assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).
Time Frame: Reporting of adverse events was required from the start of protocol therapy and until 30 days from the last administration of study drugs; up to 1 year
Population: Ineligible patients are excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Dose-Finding Level 1 CR | Dose-Finding Level 1 RT | Dose-Finding Level 2 RT | Regimen A | Regimen B | Regimen C | Regimen D
Number analyzed (Participants) | 9 | 9 | 10 | 46 | 43 | 6 | 6
Percentage of patients
  Pediatric Patients: number analyzed (Participants) | 5 | 3 | 3 | 16 | 18 | 1 | 0
  Pediatric Patients | 60 [17.06 to 100] | 66.67 [13.32 to 100] | 33.33 [0 to 86.68] | 75 [53.78 to 96.22] | 33.33 [11.56 to 55.11] | 0 [0 to 0] |
  Adult Patients: number analyzed (Participants) | 4 | 6 | 7 | 30 | 25 | 5 | 6
  Adult Patients | 75 [32.56 to 100] | 66.67 [28.95 to 100] | 57.14 [20.48 to 93.80] | 86.67 [74.50 to 98.83] | 36 [17.18 to 54.82] | 40 [0 to 82.94] | 0 [0 to 0]

10. Other Pre Specified Outcome: Relative Frequency of Actionable Mutations
Description: Descriptive statistical analyses will be provided to estimate the relative frequency of actionable mutations across the whole cohort and within more common histological subtypes, like synovial sarcoma and malignant peripheral nerve sheath tumors.
Time Frame: At diagnosis
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Prevalence of Circulating Tumor DNA (ctDNA)
Description: Descriptive analyses will be performed to summarize the prevalence of ctDNA.
Time Frame: At diagnosis
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Mean Pharmacokinetic Parameters of Doxorubicin and Pazopanib
Description: Pharmacokinetic parameters such as the clearance of doxorubicin and pazopanib will be estimated.
Time Frame: Up to 48 hours after the end of infusion
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Fludeoxyglucose F 18 (FDG) Positron Emission Tomography (PET) Maximum Standard Uptake Value (SUVmax)
Description: To evaluate change in FDG PET maximum standard uptake value (SUVmax) from baseline to Week 10 or 13 in patients with unresected tumors and to correlate this change with pathologic response and EFS.
Time Frame: From enrollment to week 10 or 13 prior to tumor resection
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Relative Risk of Failure Based on Both Standard Imaging and Pathologic Assessment
Description: To compare the rate of response by standard imaging and pathologic assessment to determine which correlates better with local tumor control, distant tumor control, event free survival, and overall survival.
Time Frame: From enrollment up to 60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Reporting of adverse events was required from the start of protocol therapy and until 30 days from the last administration of study drugs; up to 1 year
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Dose-Finding Level 1 CR | Dose-Finding Level 1 RT | Dose-Finding Level 2 RT | Regimen A | Regimen B | Regimen C | Regimen D
All-Cause Mortality (participants affected / at risk) | 1/9 | 4/9 | 3/10 | 5/46 | 9/43 | 0/6 | 2/6
Serious Adverse Events (participants affected / at risk) | 6/9 | 6/9 | 2/10 | 33/46 | 8/43 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/9 | 2/9 | 5/10 | 20/46 | 10/43 | 1/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dose-Finding Level 1 CR (N=9) | Dose-Finding Level 1 RT (N=9) | Dose-Finding Level 2 RT (N=10) | Regimen A (N=46) | Regimen B (N=43) | Regimen C (N=6) | Regimen D (N=6)
Anorexia (Metabolism and nutrition disorders) | 0/5 | 0/3 | 0/3 | 2/16 | 0/18 | 0/1 | 0/0 — Pediatric
Creatinine increased (Investigations) | 0/5 | 1/3 | 0/3 | 0/16 | 0/18 | 0/1 | 0/0 — Pediatric
Dehydration (Metabolism and nutrition disorders) | 0/5 | 0/3 | 0/3 | 2/16 | 0/18 | 0/1 | 0/0 — Pediatric
Diarrhea (Gastrointestinal disorders) | 0/5 | 0/3 | 1/3 | 0/16 | 0/18 | 0/1 | 0/0 — Pediatric
Febrile neutropenia (Blood and lymphatic system disorders) | 1/5 | 0/3 | 0/3 | 7/16 | 0/18 | 0/1 | 0/0 — Pediatric
Fever (General disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Hallucinations (Psychiatric disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Hyperkalemia (Metabolism and nutrition disorders) | 0/5 | 0/3 | 1/3 | 0/16 | 0/18 | 0/1 | 0/0 — Pediatric
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Ileus (Gastrointestinal disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Mucositis oral (Gastrointestinal disorders) | 0/5 | 0/3 | 0/3 | 3/16 | 0/18 | 0/1 | 0/0 — Pediatric
Pain (General disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Perforation bile duct (Hepatobiliary disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Sepsis (Infections and infestations) | 0/5 | 0/3 | 0/3 | 0/16 | 1/18 | 0/1 | 0/0 — Pediatric
Skin infection (Infections and infestations) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Thromboembolic event (Vascular disorders) | 1/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Vomiting (Gastrointestinal disorders) | 0/5 | 0/3 | 0/3 | 2/16 | 0/18 | 0/1 | 0/0 — Pediatric
Wound dehiscence (Injury, poisoning and procedural complications) | 0/5 | 1/3 | 0/3 | 1/16 | 1/18 | 0/1 | 0/0 — Pediatric
Wound infection (Infections and infestations) | 0/5 | 1/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Wound complication (Injury, poisoning and procedural complications) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Acute kidney injury (Renal and urinary disorders) | 0/5 | 1/3 | 0/3 | 0/16 | 0/18 | 0/1 | 0/0 — Pediatric
Alanine aminotransferase increased (Investigations) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Anemia (Blood and lymphatic system disorders) | 0/4 | 1/6 | 0/7 | 2/30 | 1/25 | 0/5 | 0 — Adult
Atrial fibrillation (Cardiac disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Atrial flutter (Cardiac disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Blood bilirubin increased (Investigations) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Blurred vision (Eye disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Chills (General disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 1/5 | 0 — Adult
Cognitive disturbance (Nervous system disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Death NOS (General disorders) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Dehydration (Metabolism and nutrition disorders) | 1/4 | 0/6 | 1/7 | 0/30 | 0/25 | 0/5 | 0 — Adult
Delirium (Psychiatric disorders) | 0/4 | 0/6 | 0/7 | 3/30 | 0/25 | 0/5 | 0 — Adult
Depression (Psychiatric disorders) | 0/4 | 0/6 | 1/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Diarrhea (Gastrointestinal disorders) | 0/4 | 0/6 | 1/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Dizziness (Nervous system disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 1/25 | 0/5 | 0 — Adult
Electrocardiogram QT corrected interval prolonged (Investigations) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Encephalopathy (Nervous system disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Esophagitis (Gastrointestinal disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Fatigue (General disorders) | 0/4 | 0/6 | 0/7 | 2/30 | 0/25 | 1/5 | 0 — Adult
Febrile neutropenia (Blood and lymphatic system disorders) | 1/4 | 0/6 | 0/7 | 11/30 | 1/25 | 0/5 | 0 — Adult
Fever (General disorders) | 0/4 | 0/6 | 0/7 | 2/30 | 2/25 | 1/5 | 0 — Adult
Gait disturbance (General disorders) | 0/4 | 1/6 | 0/7 | 0/30 | 0/25 | 0/5 | 0 — Adult
General disorders and administration site conditions - Other, specify (General disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Headache (Nervous system disorders) | 0/4 | 0/6 | 1/7 | 0/30 | 0/25 | 0/5 | 0 — Adult
Hyperglycemia (Metabolism and nutrition disorders) | 0/4 | 1/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Hypokalemia (Metabolism and nutrition disorders) | 0/4 | 1/6 | 0/7 | 2/30 | 0/25 | 0/5 | 0 — Adult
Hyponatremia (Metabolism and nutrition disorders) | 0/4 | 0/6 | 0/7 | 3/30 | 1/25 | 1/5 | 0 — Adult
Hypophosphatemia (Metabolism and nutrition disorders) | 0/4 | 0/6 | 0/7 | 3/30 | 0/25 | 1/5 | 0 — Adult
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Lymphocyte count decreased (Investigations) | 0/4 | 0/6 | 0/7 | 2/30 | 1/25 | 0/5 | 0 — Adult
Mucositis oral (Gastrointestinal disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Multi-organ failure (General disorders) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Nausea (Gastrointestinal disorders) | 1/4 | 0/6 | 0/7 | 1/30 | 0/25 | 1/5 | 0 — Adult
Neutrophil count decreased (Investigations) | 0/4 | 0/6 | 0/7 | 5/30 | 0/25 | 0/5 | 0 — Adult
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0/4 | 1/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Photophobia (Eye disorders) | 0/4 | 0/6 | 1/7 | 0/30 | 0/25 | 0/5 | 0 — Adult
Platelet count decreased (Investigations) | 0/4 | 0/6 | 0/7 | 5/30 | 0/25 | 0/5 | 0 — Adult
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0/4 | 0/6 | 0/7 | 2/30 | 0/25 | 0/5 | 0 — Adult
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Sepsis (Infections and infestations) | 0/4 | 0/6 | 0/7 | 4/30 | 1/25 | 0/5 | 0 — Adult
Sinus tachycardia (Cardiac disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0/4 | 0/6 | 1/7 | 0/30 | 0/25 | 0/5 | 0 — Adult
Skin infection (Infections and infestations) | 0/4 | 0/6 | 0/7 | 2/30 | 1/25 | 0/5 | 0 — Adult
Stroke (Nervous system disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Syncope (Nervous system disorders) | 1/4 | 0/6 | 0/7 | 0/30 | 0/25 | 0/5 | 0 — Adult
Thromboembolic event (Vascular disorders) | 1/4 | 1/6 | 0/7 | 4/30 | 0/25 | 0/5 | 0 — Adult
Upper respiratory infection (Infections and infestations) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Urinary tract infection (Infections and infestations) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Uterine hemorrhage (Reproductive system and breast disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Vomiting (Gastrointestinal disorders) | 1/4 | 0/6 | 1/7 | 2/30 | 0/25 | 0/5 | 0 — Adult
Wound dehiscence (Injury, poisoning and procedural complications) | 2/4 | 0/6 | 0/7 | 4/30 | 0/25 | 0/5 | 0 — Adult
Wound infection (Infections and infestations) | 1/4 | 3/6 | 1/7 | 1/30 | 1/25 | 0/5 | 0 — Adult
White blood cell decreased (Investigations) | 0/4 | 0/6 | 0/7 | 8/30 | 0/25 | 0/5 | 0 — Adult
Ejection fraction decreased (Investigations) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Wound complication (Injury, poisoning and procedural complications) | 0/4 | 0/6 | 0/7 | 2/30 | 1/25 | 0/5 | 0 — Adult
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Dermatitis radiation (Injury, poisoning and procedural complications) | 0/4 | 0/6 | 1/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Lung infection (Infections and infestations) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Soft tissue infection (Infections and infestations) | 0/4 | 1/6 | 0/7 | 0/30 | 0/25 | 0/5 | 0 — Adult
Non-cardiac chest pain (General disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Device related infection (Infections and infestations) | 0/4 | 0/6 | 0/7 | 1/30 | 1/25 | 0/5 | 0 — Adult
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dose-Finding Level 1 CR (N=9) | Dose-Finding Level 1 RT (N=9) | Dose-Finding Level 2 RT (N=10) | Regimen A (N=46) | Regimen B (N=43) | Regimen C (N=6) | Regimen D (N=6)
Alanine aminotransferase increased (Investigations) | 1/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Cardiac disorders - Other, specify (Cardiac disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Hypertension (Vascular disorders) | 1/5 | 0/3 | 0/3 | 0/16 | 0/18 | 0/1 | 0/0 — Pediatric
Lymphocyte count decreased (Investigations) | 1/5 | 0/3 | 0/3 | 3/16 | 2/18 | 0/1 | 0/0 — Pediatric
Neutrophil count decreased (Investigations) | 1/5 | 0/3 | 0/3 | 4/16 | 5/18 | 0/1 | 0/0 — Pediatric
Platelet count decreased (Investigations) | 0/5 | 0/3 | 0/3 | 3/16 | 2/18 | 0/1 | 0/0 — Pediatric
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Wound dehiscence (Injury, poisoning and procedural complications) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
White blood cell decreased (Investigations) | 1/5 | 0/3 | 0/3 | 4/16 | 3/18 | 0/1 | 0/0 — Pediatric
Wound complication (Injury, poisoning and procedural complications) | 1/5 | 0/3 | 0/3 | 0/16 | 0/18 | 0/1 | 0/0 — Pediatric
Localized edema (General disorders) | 0/5 | 0/3 | 0/3 | 1/16 | 0/18 | 0/1 | 0/0 — Pediatric
Alanine aminotransferase increased (Investigations) | 0/4 | 0/6 | 1/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Anemia (Blood and lymphatic system disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Aspartate aminotransferase increased (Investigations) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Fatigue (General disorders) | 0/4 | 1/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Febrile neutropenia (Blood and lymphatic system disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 2/25 | 0/5 | 0 — Adult
Hyperkalemia (Metabolism and nutrition disorders) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Hyperphosphatemia (Metabolism and nutrition disorders) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Hypertension (Vascular disorders) | 0/4 | 1/6 | 1/7 | 0/30 | 0/25 | 1/5 | 0 — Adult
Hypokalemia (Metabolism and nutrition disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Hypotension (Vascular disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Infections and infestations - Other, specify (Infections and infestations) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Lipase increased (Investigations) | 0/4 | 0/6 | 0/7 | 0/30 | 1/25 | 0/5 | 0 — Adult
Lymphocyte count decreased (Investigations) | 1/4 | 0/6 | 1/7 | 2/30 | 3/25 | 0/5 | 0 — Adult
Neutrophil count decreased (Investigations) | 1/4 | 0/6 | 0/7 | 10/30 | 2/25 | 0/5 | 0 — Adult
Platelet count decreased (Investigations) | 0/4 | 0/6 | 0/7 | 5/30 | 2/25 | 0/5 | 0 — Adult
Urinary tract infection (Infections and infestations) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
Wound dehiscence (Injury, poisoning and procedural complications) | 0/4 | 0/6 | 2/7 | 0/30 | 0/25 | 0/5 | 0 — Adult
Wound infection (Infections and infestations) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult
White blood cell decreased (Investigations) | 1/4 | 0/6 | 0/7 | 6/30 | 2/25 | 0/5 | 0 — Adult
Wound complication (Injury, poisoning and procedural complications) | 0/4 | 0/6 | 0/7 | 0/30 | 0/25 | 1/5 | 0 — Adult
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0/4 | 0/6 | 0/7 | 1/30 | 0/25 | 0/5 | 0 — Adult

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT02180867/Prot_SAP_001.pdf